CLINICAL TRIAL: NCT00585572
Title: University of Wisconsin-Madison: Wisconsin Brain Donor Program (WBDP)
Brief Title: Wisconsin Brain Donor Program
Acronym: WBDP
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: University of Washington (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: H-2010-0037; H-2010-0037 (Other: Minimal Risk Research IRB); 2014-1484 (Other: Minimal Risk Research IRB); A534255 (Other: UW Madison); GERIATRICS AND ADULT (Other: UW Madison); 2RF1AG027161-11A1 (NIH); 1P30AG062715-01 (NIH)
Record Dates: First submitted 2007-12-26; First posted 2008-01-03 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment
Keywords: Normal Tissues/Brains; Alzheimer; Motor Neuron Disease; Dementia; Healthy Control Volunteers; Populations At Risk; MCI
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Motor Neuron Disease; Dementia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Brain tissue, blood, cerebrospinal fluid, spinal cord, peripheral nerves, and skeletal muscles, central/peripheral nervous tissue, as well as skeletal muscle tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Wisconsin Brain Donor Program (WBDP) stores brain and other tissues/samples (e.g. blood and CSF) from deceased individuals who have participated in longitudinal research studies, as well as other select participants. These individuals have donated their tissues in order to aid scientific research. Through the collection of central and peripheral nervous tissues as well as (in select cases) skeletal muscle tissue, the WBDP strives to advance the knowledge of diseases of memory disorders, such as Alzheimer's Disease. Brain donations are needed from healthy individuals, as well as those affected by diseases of the nervous system.

DETAILED DESCRIPTION:
The Wisconsin Brain Donor Program (WBDP) of the University of Wisconsin-Madison School of Medicine and Public Health is considered an investigator-initiated project. It was first established in 1995 to promote teaching and research in neurodegenerative diseases. In 2009 the WBDP aligned itself with the research goals of the Wisconsin Alzheimer's Disease Research Center (Wisconsin ADRC) in order to more effectively serve the research community. As a result, the WBDP is part of a nationwide network of ADC/ADRC's (Alzheimer's Disease Centers/Alzheimer's Disease Research Centers), funded by the National Institute on Aging that exists to promote research on neurodegenerative diseases. However, the WBDP operates as an independent research program under the direction of the WBDP and Wisconsin ADRC Principal Investigators.

The WBDP provides approved researchers access to indefinitely-stored postmortem brain tissues and post-mortem biospecimens (subject to the availability of remaining stock). Postmortem biospecimens also include CSF and whole blood.

The WBDP staff promotes and educates the lay community on the importance of brain donation.

Goal/Objectives The overall goal of the WBDP is to function as a useful brain tissue and biospecimen repository by distributing these materials to approved researchers studying neurodegenerative diseases, particularly Alzheimer's disease (AD).

To achieve this goal, the WBDP has adopted the following overall objectives:

1. To serve as the tissue and biospecimen repository for the Wisconsin ADRC and Wisconsin ADRC-affiliated studies. In this role, the WBDP will support collaborative research by providing postmortem tissues, biospecimens, and genetic/genomic data for AD and other neurodegenerative illnesses to approved researchers, whether at the University of Wisconsin-Madison or other approved institutions. The investigators will also promote data and sample sharing with ADRC Clinical Core, WRAP, and ADRC-affiliated studies such as ADNI, DOD-ADNI, and ADNI Brain Bank.
2. To establish a registered group of individuals who intend to donate their brain tissue and biospecimens after death for neurodegenerative-disease related research (the WBDP Registry).
3. To oversee all aspects of brain tissue and biospecimen collection and management (their procurement, indefinite storage, and distribution to approved researchers).
4. To collaborate with the National Alzheimer's Coordinating Center (NACC), the National Centralized Repository for Alzheimer's Disease and Related Dementias (NCRAD) and similar organizations, by providing coded biologic samples and data, inclusive of genetic data, in order to further AD research.

Due to the nature of this study, no specific number of subjects is being proposed. This will be an ongoing brain donation registry until funding is not renewed.

ELIGIBILITY:
Inclusion Criteria:

* Is aged 18 years or older
* Falls into one of the following categories:

  * Current or previous study participants involved in the ADRC Clinical Core, WRAP study, or other select ADRC-affiliated studies, or donors of special circumstance, including healthy controls, if approved on a case-by-case basis by the WBDP PI. Please note, ADRC-affiliated studies are not inclusive of ADRC-affiliated industry-sponsored studies.
  * Is a parent of either an ADRC Clinical Core or WRAP study participant, or is a spouse of a WRAP study participant.

Exclusion Criteria:

* VA research subjects
* Subjects with a medical condition/disease that would exclude them from the spectrum of utility/interest to researchers as determined by a WBDP Neuropathologist:

  1. Persons with Hepatitis B or C
  2. Severe Traumatic Brain Injury
  3. Positive CJD diagnosis
  4. Persons with HIV/AIDS
  5. Persons with brain tumors or blood clots that affect neurologic status, therefore creating a problem between diagnosing AD status and healthy status
  6. Cancer that has metastasized to the brain
  7. Radiation treatment to the head
  8. Other infectious diseases that would be hazardous to staff handling the tissue
  9. Prolonged ventilator dependency prior to death as determined by the Neuropathologist
* Subjects who lack capacity to provide informed consent with no activated Power of Attorney (POA) for Healthcare, activated POA for Research, or legal guardianship (if not near death), or (if at or near death) have no spouse, parent, relative or friend willing/able to complete consent and other donation paperwork.
* Subjects who otherwise have incomplete history or incomplete donation paperwork before a recovery can begin.
* Subjects younger than 18 years of age.
* An expected post-mortem interval (PMI) of greater than 16 hours for non-ADRC or non-WRAP participants. PMI is the time between death and the anticipated time of brain removal at autopsy. Families and recovery agencies are made aware of this time constraint when consenting for the recovery process. If a patient becomes ineligible due to PMI, the family and funeral home will be notified immediately. Diversions from this exclusion can be made by a WBDP PI or Co-PI.
* Medical conditions that would put researchers at risk.
* Other contingencies, as determined by the PI, that make enrollment impractical or unsafe.

Note: It is anticipated, based upon the younger age of our study cohorts, that significant time may pass between WBDP registration and actual donation. The inclusion/exclusion criteria will be reviewed and applied at time of donation. As a result, donated tissue found to be unsuitable may be removed from the post-mortem tissue and biosamples collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants agree to autopsy and brain/tissue/sample donation for research purposes only.
Sampling Method: Non-Probability Sample
Enrollment: 9999 (Estimated)
Dates: Start 2007-03 (Actual); Primary Completion 2050-08 (Estimated); Study Completion 2050-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shahriar Salamat, MD PHD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Madison, Madison, Wisconsin, United States